CLINICAL TRIAL: NCT04716114
Title: A Phase 3, Open-Label, Multicenter, Randomized Study of SKLB1028 Versus Salvage Chemotherapy in Patients With FLT3-mutated Acute Myeloid Leukemia Refractory to or Relapsed After First-line Treatment（ALIVE）
Brief Title: A Study of SKLB1028 Versus Salvage Chemotherapy in Patients With Relapsed or Refractory (R/R) AML With FLT3-Mutated
Acronym: ALIVE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA114-CSP-003
Record Dates: First submitted 2020-12-31; First posted 2021-01-20 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: monotherapy; SKLB1028
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — SKLB1028; Cytarabine; Azacitidine; fludarabine; Homoharringtonine; Aclarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKLB1028 (Experimental): Subjects will receive 150 mg orally twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: SKLB1028
- Salvage Chemotherapy (Active Comparator): Chemotherapy will be given in 28-day cycles. Subjects on low-dose cytarabine (LoDAC) will receive 10 to 20 mg of cytarabine twice daily by subcutaneous (SC) or intravenous (IV) injections for 7 to 14 days.
  Subjects on azacitidine will receive 75 mg/m^2 daily by SC or IV, for 5 to 7 days.
  Subjects on homoharringtonine (HHT), cytarabine and aclarubicin (HAA) will receive 2 mg/m^2 of HHT by IV, for 7 days (day 1 to 7) (or HHT 2 mg/m^2, twice daily, day 1 to 3); 100~200 mg/m^2 of cytarabine by IV for 7 days (day 1~7) and 20 mg/d of aclarubicin by IV for 7 days (day 1 to 7).
  Subjects on fludarabine, cytarabine and granulocyte colony-stimulating factor (G-CSF) (FLAG) will receive 30 mg/m^2 of fludarabine daily by IV for 5 days (day 2 to 6), 1000~2000 mg/m2 of cytarabine daily by IV for 5 days (day 2 to 6), and 300 g/m^2 of G-CSF daily by SC or IV for 5 days (days 1 to 5). After completion of chemotherapy, G-CSF will be administered continually until ANC>0.5 x 10^9 / L.
  Interventions: Drug: Salvage Chemotherapy

INTERVENTIONS:
Drug: SKLB1028 — SKLB1028 will be administered by oral capsules, 150 mg twice daily (BID).
  Arms: SKLB1028
Drug: Salvage Chemotherapy — Low-dose cytarabine (LoDAC); azacytidine; homoharringtonine (HHT), cytarabine and aclarubicin (HAA) or fludarabine, cytarabine and granulocyte colony-stimulating factor (FLAG) will be administered by subcutaneous (SC) and/or intravenous (IV) injections.
  Other Names: cytarabine, azacytidine, fludarabine, homoharringtonine, aclarubicin
  Arms: Salvage Chemotherapy

SUMMARY:
This is a randomized，multicenter, open-label Phase III, clinical study to confirm the efficacy and safety of SKLB1028 in patients with relapsed or refractory(R/R) FLT3-Mutated Acute Myeloid Leukemia（AML）compared to salvage chemotherapy.

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a 2:1 ratio to receive SKLB1028 or salvage chemotherapy. Subjects will enter the screening period up to 14 days before the start of treatment. Prior to randomization, a salvage chemotherapy regimen will be pre-selected for each subject. Options will include low-dose cytarabine (LoDAC), azacitidine, homoharringtonine (HHT), cytarabine and aclarubicin (HAA) or fludarabine, cytarabine and granulocyte colony-stimulating factor (FLAG). The randomization will be stratified by indications and intensity of pre-selected salvage chemotherapy.

Subjects will be orally administrated SKLB1028 twice daily over continuous 28-day cycles . Subjects in the salvage chemotherapy group will receive chemotherapy as required by the guidelines. Subjects receiving SKLB1028, LoDAC, or azacytidine will continue to receive the treatment until a treatment discontinuation criterion is met. Subjects receiving HAA or FLAG will take 1 cycle of therapy and will be assessed for response after the 1st cycle. After the efficacy evaluation, the subject may receive a second cycle of chemotherapy at the investigator's discretion. will receive the second cycle of chemotherapy.

Subjects who have a donor identified and with complete remission after treatment may undergo hematopoietic stem cell transplant (HSCT) without leaving the study. Subjects in the salvage chemotherapy group who withdrew due to non-response to treatment or disease progression, could switch to SKLB1028 if SKLB1028 will likely benefit the patient at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed the informed consent form.
2. Age≥18 years old, no gender limitation.
3. Patient has a diagnosis of primary AML or AML secondary to myelodysplastic syndrome (MDS) as determined by pathological and morphological results, according to World Health Organization (WHO) 2016 classification.
4. Patient is refractory to or relapsed after first-line AML therapy (with or without HSCT).

   1. Refractory to first-line AML treatment is defined as: the patient did not achieve complete remission/complete remission with incomplete hematologic recovery/complete remission with incomplete platelet recovery (CR/CRi/CRp) under initial therapy. A patient eligible for standard therapy must receive at least 1 cycle of an anthracycline containing induction therapy in the standard dose for the selected induction regimen. A patient not eligible for standard therapy must have received at least 1 complete block of induction therapy seen as the optimum choice of therapy to induce remission for this patient as per investigator's assessment.
   2. Early relapse after first-line AML therapy is defined as: the patients achieved CR/CRi/CRp after first-line treatment, and relapsed within 6 months with hematological relapse.
   3. Advanced relapse after first-line AML therapy is defined as: the patients achieved CR/CRi/CRp after first-line treatment and relapsed after 6 months with hematological relapse;
5. Patient is positive for FLT3 mutation in bone marrow or whole blood.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Patient is eligible for pre-selected salvage chemotherapy according to investigator assessment.
8. Patient must meet the following criteria as indicated on the clinical laboratory tests:

   1. Serum aspartate aminotransferase and alanine aminotransferase ≤ 3.0 x upper limit of normal (ULN);
   2. Serum total bilirubin ≤ 1.5 x ULN;
   3. Serum creatinine ≤ 3.0 x ULN or an estimated glomerular filtration rate of > 30 mL/min.
9. Patient is suitable for oral administration of the study drug.
10. Female or male patient of childbearing age agree to take effective non-drug contraception from the date of signing an informed consent to 180 days after the last dose and will not donate sperm or eggs.

Exclusion Criteria:

1. Patient was diagnosed as acute promyelocytic leukemia (APL), or BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
2. Patient has AML secondary to prior chemotherapy for other neoplasms (except for MDS).
3. AML with central nervous system (CNS) involvement (defined as highly suspected CNS involvement with clinical symptoms supported by imaging evidence).
4. Refractory hypokalemia or hypomagnesemia that is difficult to be corrected by symptomatic treatment and has recurred in the past.
5. Patient is currently suffering from clinically significant graft-versus-host disease (GVHD) or receiving systemic cortisol hormone therapy for GVHD.
6. Patient has been previously diagnosed with another malignancy (except in the following cases: disease-free for at least 5 years; Patients with treated nonmelanoma skin cancer, breast in situ carcinoma or cervical intraepithelial neoplasia [regardless of disease status]; Localized prostate cancer with no recurrence or progression that is expected to be cured after treatment, such as radiotherapy or surgery)
7. Patient has clinically significant abnormality of coagulation profile, such as disseminated intravascular coagulation (DIC), hemophilia A, hemophilia B, and von Willebrand disease.
8. Patient has had major surgery within 4 weeks prior to the study (the definition of major surgery was based on the level 3 and level 4 surgeries stipulated in the Management Measures for Clinical Application of Medical Technology), or has not fully recovered from any previous invasive operation.
9. Patient has radiation therapy within 4 weeks before the first study dose.
10. Patient has congestive heart failure New York Heart Association (NYHA) class 3 or 4 or patient with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 1 month before study entry results in a left ventricular ejection fraction that is ≥ 45%.
11. Patient has bradycardia and heart rate is less than 50 beats/min, except for pacemaker user.
12. Patients with mean value of triplicate Fridericia-corrected QT interval (QTcF) in the screening period, male > 450 ms, female > 470 ms.
13. Patients with diagnosed or suspected long QT syndrome at screening (including a family history of long QT syndrome).
14. Patients with second degree (Mobitz II) or third degree atrioventricular block disease (except for patients who use the pacemaker).
15. Patients with uncontrolled angina or myocardial infarction in 6 months before screening.
16. Patient has a complete left bundle branch block during screening.
17. Patients with new clinically significant arrhythmias (except for sinus tachycardia caused by anemia, infection and AML) or patients with previous arrhythmias that require long-term use of drugs with QT-prolonging effects.
18. Patient has an active uncontrolled infection.
19. Patients are hepatitis B surface antigen-positive or have a history of hepatitis B, with HBV-DNA ≥2000 IU/mL in the past 3 months; Patients are hep
20. Patients with positive anti-human immunodeficiency virus antibodies or anti-Treponema pallidum specific antibodies.
21. Patient has cytotoxic chemotherapy drugs <2 weeks, or non-cytotoxic drugs <5 half-lives prior to the first study dose (except hydroxyurea and other treatments used to control hyperleucocytosis).
22. Patients have taken CYP 2C8 and CYP 3A4 strong inducers or inhibitors within 2 weeks prior to the first study dose.
23. Patients have previously received other FLT3 inhibitors (Gilteritinib, Quizatinib, Crenolanib, etc.), except for sorafenib.
24. Pregnant (blood pregnancy test positive in screening period) and lactating Female.
25. Patients are not suitable for the study in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Interim analysis: CR/CRh rate in the experimental group. | up to 4 years.
  The complete remission and complete remission with partial hematological recovery (CR/CRh) rate was defined as the number of subjects who achieved either CR or CRh divided by the number of subjects in the response analysis set (RAS).
The final analysis: Overall Survival(OS) | up to 4 years.
  Overall survival was defined as the time from the date of randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Key secondary end point: Event-Free Survival (EFS). | up to 4 years.
  EFS was defined as the time from randomization until treatment failure (Composite complete remission (CRc) or partial remission (PR) were not reached within 4 cycles), relapse (excluding relapse after PR), or death from any cause, whichever occurs first.
Duration of remission (DOR). | up to 4 years.
  Duration of remission included duration of composite complete remission (CRc), duration of complete remission (CR)/ complete remission with partial hematologic recovery (CRh), duration of CRh, duration of CR and duration of response (CRc + partial remission (PR).
Duration of Leukemia-Free Survival (LFS) | up to 4 years.
  The LFS was defined as the time from the date of first CR until the date of documented relapse (excluding relapse from PR) or death for participants who achieved CR (relapse date or death date - first CR disease assessment date + 1).
Composite complete remission rate | up to 4 years.
  CR rate was defined as the number of participants who achieved the best response of CR divided by the number of participants in the analysis population.
Time to CR(TTR) | up to 4 years.
  Time to CR(TTR) is defined as the time from the date of randomization until the date of is defined as the time from the date of randomization until the date of CR
Transplantation rate | up to 4 years.
  Transplantation rate is defined as the percentage of participants undergoing hematopoietic stem cell transplant (HSCT).
Transfusion conversion rate and transfusion-Independence rate. | up to 4 years.
  Transfusion conversion rate is defined as subjects whose baseline transfusion-dependent (TD, received red blood cell or platelet transfusion within 28 days prior to C1D1) to non-transfusion-dependent (Transfusion-Independence, TI, ≥56 days without red blood cell or platelet transfusion) Proportion; non-transfusion dependent maintenance rate is defined as the proportion of subjects who maintain TI status during the trial period of baseline non-transfusion dependent (TI) subjects.
Safety assessed by adverse events. | up to 4 years.
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment.
Population pharmacokinetic of SKLB1028 | Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1: predose. A cycle is 28 days.
  Observed trough concentration (Ctrough)

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital of Sichuan University, Chengdu, Sichuan, China